CLINICAL TRIAL: NCT00829504
Title: The Relative Bioavailability Study of Two Ropinirole 0.25 mg Tablets Under Fasting Conditions.
Brief Title: Ropinirole 0.25 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 10436008
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2009-09-11 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — ropinirole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Ropinirole HCl 0.25 mg Tablets
- 2 (Active Comparator)
  Interventions: Drug: Requip® 0.25 mg Tablets

INTERVENTIONS:
Drug: Ropinirole HCl 0.25 mg Tablets — 1 x 0.25 mg
  Arms: 1
Drug: Requip® 0.25 mg Tablets — 1 x 0.25 mg
  Arms: 2

SUMMARY:
The objective of this study was to compare the relative bioavailability of the test formulation of Ropinirole (TEVA Pharmaceuticals USA) with already marketed reference of Requip® (Manufactured by SmithKline Beecham Pharmaceuticals for GlaxoSmithKline) under fasting conditions in healthy, non-smoking, adult subjects.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Healthy (physical exam, laboratory tests, medical history and ECG), non-smoker males and/or females who were between 18 and 45 years old

Exclusion Criteria:

* If female, pregnant, lactating or likely to become pregnant during this study.
* History of allergy or sensitivity to ropinirole or other dopamine agonists (e.g. Corolpam®, Dostinex®, Mirapex®, Permax®, Symmetrel®) or history of any drug hypersensitivity of intolerance which, in the opinion of the Investigator, would compromise the safety of the subject or the study.
* History of dizziness, lightheadedness or fainting upon standing.
* Significant history or current evidence of chronic infectious disease, system disorders, organ dysfunction, hyper/hypotension, arrythmia, tachycardia, seizure disorder or glaucoma.
* Presence of gastrointestinal disease or history of malabsorption within the last year.
* History of psychiatric disorders occuring within the last two years that required hospitalization or medication.
* Presence of a medical condition requiring regular treatment with prescription drugs.
* Use of pharmacologic agents known to significantly induce or inhibit drug-metabolizing enzymes within 30 days prior to dosing.
* Receipt of any drug as part of a research study within 30 days prior to dosing.
* Drug or alcohol addiction requiring treatment in the past 12 months.
* Donation or significant loss of whole blood (480 ml or more) within 30 days or plasma within the past 14 days prior to dosing.
* Positive test results for HIV, Hepatitis B surface antigen or Hepatitis C antibody.
* Positive test results for drugs of abuse at screening.
* Tobacco user within 90 days of the first study date.
* Unable, or unwilling to tolerate multiple venipunctures.
* Difficulty fasting or eating the standard meals that will be provided.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2004-10; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soran Hong, M.D., Principal Investigator — Novum Pharmaceuticals Research Services
Locations (1):
- Novum Pharmaceutical Research Services, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Test (Ropinirole HCl) First: 0.25 mg Ropinirole HCl Tablets test product dosed in first period followed by 0.25 mg Requip® Tablets reference product dosed in the second period.
- Reference (Requip®) First: 0.25 mg Requip® Tablets reference product dosed in first period followed by 0.25 mg Ropinirole HCl Tablets test product dosed in the second period.
Period: First Intervention
Arm/Group | Test (Ropinirole HCl) First | Reference (Requip®) First
Started | 22 | 22
Completed | 21 | 22
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Washout of 7 Days
Arm/Group | Test (Ropinirole HCl) First | Reference (Requip®) First
Started | 21 | 22
Completed | 20 | 22
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention
Arm/Group | Test (Ropinirole HCl) First | Reference (Requip®) First
Started | 20 | 22
Completed | 19 | 22
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test (Ropinirole HCl) First | Reference (Requip®) First | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 17 | 12 | 29
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 13 | 17 | 30
  White | 0 | 1 | 1
  Hispanic | 9 | 4 | 13
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration of Drug Substance in Plasma)
Description: Bioequivalence based on Cmax.
Time Frame: Blood samples collected over a 24 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Test (Ropinirole HCl): 0.25 mg Ropinirole HCl Tablets test product dosed in either period.
- Reference (Requip®): 0.25 mg Requip® Tablets reference product dosed in either period.
Arm/Group | Test (Ropinirole HCl) | Reference (Requip®)
Number analyzed (Participants) | 40 | 40
pg/mL | 552.1 (219.01) | 546.5 (205.72)
Statistical Analysis 1: Comparison: Test (Ropinirole HCl) vs Reference (Requip®); Test type: Non-Inferiority or Equivalence — The ANOVA model was utilized in comparing the effects between the test and reference products. Differences were declared statistically significant at the 5% level (p<0.05); Ratio of the T/R geometric mean x 100 = 100.16, 90% CI [95.5 to 105.04] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference and test product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t (Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on AUC0-t.
Time Frame: Blood samples collected over a 24 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Test (Ropinirole HCl) | Reference (Requip®)
Number analyzed (Participants) | 40 | 40
pg*h/mL | 4190.92 (2290.13) | 4062.99 (2073.39)
Statistical Analysis 1: Comparison: Test (Ropinirole HCl) vs Reference (Requip®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 101.76, 90% CI [95.45 to 108.49] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf (Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on AUC0-inf.
Time Frame: Blood samples collected over a 24 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Test (Ropinirole HCl) | Reference (Requip®)
Number analyzed (Participants) | 40 | 40
pg*h/mL | 4469 (2561.37) | 4305.88 (2283.55)
Statistical Analysis 1: Comparison: Test (Ropinirole HCl) vs Reference (Requip®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 102.1, 90% CI [95.64 to 109] — [estimate comment as in outcome 1, analysis 1]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.